CLINICAL TRIAL: NCT05846945
Title: Effect of Threshold Inspiratory Trainer Versus Trigger Sensitivity Adjustment on Weaning From Mechanical Ventilation
Brief Title: Threshold Inspiratory Trainer Versus Trigger Sensitivity Adjustment on Weaning From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ICU2022
Record Dates: First submitted 2022-12-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMT group (Active Comparator): Training by inspiratory muscle device plus chest physiotherapy
  Interventions: Other: Threshold inspiratory muscle trainer device; Other: Chest physiotherapy
- TS group (Active Comparator): Adjusting trigger sensitivity of the mechanical ventilator to the lowest pressure tolerated plus chest physiotherapy
  Interventions: Other: Adjusting mechanical ventilator trigger sensitivity; Other: Chest physiotherapy
- PT group (Sham Comparator): Routine chest physiotherapy
  Interventions: Other: Chest physiotherapy

INTERVENTIONS:
Other: Threshold inspiratory muscle trainer device — The threshold inspiratory muscle trainer (IMT) device offers resistance to respiration through the spring-loaded valve.
  Arms: IMT group
Other: Adjusting mechanical ventilator trigger sensitivity — modifying the mechanical ventilator trigger sensitivity so that patients can only initiate inspiratory flow by producing more negative intrathoracic pressure
  Arms: TS group
Other: Chest physiotherapy — Conventional chest physiotherapy

SUMMARY:
Ninety adult patients from both gender, with acute respiratory failure, intubated and mechanically ventilated. Their ages ranged from 50 to 70 years. They were selected from Intensive Care Unit (ICU), Department of Chest Diseases, Cairo University Hospitals. They have randomly assigned into three equal groups. Group (A): trained by threshold IMT device plus routine physical therapy. Group (B): trained by adjusting MV trigger sensitivity plus routine physical therapy. Group (C): only received routine physical therapy. (Negative inspiratory force NIF, arterial blood gases, P/F ration, respiratory rate RR, tidal volume VT, and rapid shallow breathing index RSBI) were measured before the study and at the end of the study (just before weaning for successfully weaned patients, or on the 10 day of intervention for failed weaning patients).

ELIGIBILITY:
Inclusion Criteria:

* Their age ranged from 50-70 years.
* The patients were diagnosed with acute respiratory failure duo to COPD exacerbation and need mechanical ventilation support for more than 48 hours.
* They were vitally stable and can tolerate pressure support
* PEEP less than 8Cm H2O , SpO2 more than 90).
* All patients were conscious and responded to verbal command.

Exclusion Criteria:

* Unstable hemodynamics,
* unstable neurological problems,
* lack of attention and cooperation
* skipping more than five training sessions.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
partial pressure of oxygen(PaO2) | change from baseline at one week
  arterial blood sample was taken and examined thePao2
partial pressure of carbon dioxide(PaCO2) | change from baseline at one week
  arterial blood sample was taken and examined the PaCO2

SECONDARY OUTCOMES:
Respiratory rate (RR) | change from baseline at one week
  Number of respiratory cycles per minute
tidal volume (TV) | change from baseline at one week
  volume of air inspired in quiet breathing

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No